CLINICAL TRIAL: NCT05727150
Title: Reliability and Versatility of Supraclavicular Artery Flap in Reconstruction of Head and Neck Soft Tissue Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmad Ahmad Albadry, Resident,Plastic Surgery Department,Principal investigator, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-01-03
Record Dates: First submitted 2023-01-22; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Reconstruction of Head Soft Tissue Defects; Reconstruction of Neck Soft Tissue Defects

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient operated by Supraclavicular Artery flap for Reconstruction (Experimental): Supraclavicular artery flap will be used for reconstruction
  Interventions: Procedure: Reconstruction of Soft tissue defects of head and neck by Supraclavicular artery flap

INTERVENTIONS:
Procedure: Reconstruction of Soft tissue defects of head and neck by Supraclavicular artery flap — Supraclavicular artery flap will be used in the reconstruction of traumatic and non-traumatic defects of head and neck.Flap harvesting and reconstruction will be performed under general anesthesia. The defect dimensions are measured and the superficial landmarks for the supraclavicular artery are drawn .The flap will be used as island flap, transposed or interpolated flap depending on the arc of rotation needed to achieve flap inset without tension and flap elevation proceeds from lateral to medial.The flap is rotated and inset into the defect

SUMMARY:
This is a case series study conducted at plastic surgery department Sohag University including 20 patients The aim of this thesis is to evaluate reliability and versatility of Supraclavicular artery flap in the reconstruction of traumatic and non-traumatic defects of head and neck.With adequate documentation of functional, aesthetic outcome and patient satisfaction through; clinical examination , photographic documentation and doctor and patient satisfaction charts

ELIGIBILITY:
Inclusion Criteria:

* Patients with head and neck soft tissue defect either traumatic or non-traumatic
* Available healthy donor site

Exclusion Criteria:

* Trauma or conditions affecting donor site or with possible compromise of vascular pedicle.
* Patients with a major uncontrollable medical illness, chronic heavy smokers.

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Flap Success | 6 month post-surgery
  The flap success will be measured by percentage of patients in which there is flap survival versus percentage of patient with flap necrosis
Flap complications | 6 months post-surgery
  assessment of flap complication will be assessed by percentage of patients in which there is flap dehiscence , flap infection and flap necrosis
patients satisfaction as regard flap color match | 6 months post-surgery
  patient satisfaction as will be assessed with questionnaire
patients satisfaction as regard flap texture match | 6 months post-surgery
  patient satisfaction as will be assessed with questionnaire

SECONDARY OUTCOMES:
Possible flap lengths | 6 months post-surgery
  The achieved flap length will be measured in centimeters
Possible flap widths | 6 months post-surgery
  The achieved flap width will be measured in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad A Albadry, Principal Investigator — Sohag University
Locations (1):
- Sohag Faculty of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided